CLINICAL TRIAL: NCT03478228
Title: Balance Among People With Fall-related Wrist Fractures and Effects of Sensory Training
Brief Title: Multi-Sensory Training and Wrist Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Landspitali University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2013 16 ÓB/eí
Record Dates: First submitted 2018-03-19; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Postural Balance
Keywords: fracture; rehabilitation; wrist; sensation; exercise
MeSH Terms: conditions — Fractures, Bone; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Multi-Sensory Training (MST) (Experimental): Multi-Sensory Training. 6 treatment sessions, supervised by a physiotherapist, during a 3 months training period, and a written exercise program that is to be performed daily at home. The participants keep a home exercise diary during the training period.
  Interventions: Other: Multi-Sensory Training
- Wrist Stabilisation Training (WT) (Active Comparator): Wrist Stabilisation Training. 6 treatment sessions, supervised by a physiotherapist, during a 3 months training period, and a written exercise program that is to be performed daily at home. The participants keep a home exercise diary during the training period.
  Interventions: Other: Multi-Sensory Training

INTERVENTIONS:
Other: Multi-Sensory Training
  Other Names: Wrist Stabilisation Training

SUMMARY:
The aim of the study is to investigate whether individuals with fall-related wrist fractures have impaired posterior control, reduced proprioception in their lower limbs and/or vestibular asymmetry compared with those who have not fallen and sustained a fracture. Secondly to investigate the effects of a new balance training method, directed at the sensory systems and training of fall-preventive movements on postural control and how it impacts the function of the sensory systems. Postural instability falls and fractures form one of the major problems associated with ageing. An association of vestibular- asymmetry with falls and fractures has been found and reduced vibration sensation in the lower limbs has been connected with imbalance. Wrist fractures are often precursor to the more serious hip fractures, which often result in decreased quality of life, even death and are costly for the society. Subjects will be individuals 50-75 years of age having sustained a fall-related wrist fracture. Measurements of sensory functions, postural control and functional ability will be conducted before and after balance training. Confidence in daily activities and self-perceived dizziness handicap will be obtained with questionnaires. The same evaluations will be performed on age and gender matched individuals without previous history of fall-related wrist fractures. This research might reveal the presence and frequency of vestibular asymmetry or/and other age related degenerative changes in the sensory systems, which decrease stability and increase the risk of falls and fractures. It could show preventive effects of specific balance training on fall risk, and thus increase quality of life of the individuals, improve healthcare services and decrease costs associated with falls and fractures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50-75 years
* Sustained a fall-related wrist fracture
* Mentally and physically able to understand and undergo the study measurements and training.

  * Able to walk 30 metres unsupported or with an aid of a stick/crutch
  * Able to stand unsupported for ten minutes
  * Normal corrective vision
* Have signed an informed consent for participation in the study

Exclusion Criteria:

Confirmed diagnosis of degenerative Central Nervous System (CNS) diseases, such as Parkinson, Alzheimer and other diseases impairing mobility and cognitive function and hence precluding participation in the study.

More detailed exclusions criteria:

* Previous history of stroke
* Parkinson
* MS
* Multisystem atrophy
* Motor neuron disease
* Dementia, decline of cognitive function
* Serious mental illness
* Amputation in lower limbs
* Epilepsy on medical treatment

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-05-15 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
Sensory Organization Test (SOT) | 14 weeks
  Balance measurement

CONTACTS AND LOCATIONS:
Overall Officials: Palmi V Jonsson, MD, Study Chair — Landspitali National University Hospital
Locations (1):
- University of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No